CLINICAL TRIAL: NCT01006564
Title: Multifunctional MR for Radiotherapy Planning in Prostate Cancer
Brief Title: Multifunctional Magnetic Resonance (MR) for Radiotherapy Planning in Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Dr Nandita deSouza, Institute of Cancer Research
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: CCR3121
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
Keywords: Magnetic Resonance Imaging; Prostate Cancer; Magnetic Resonance Spectroscopy; Radiotherapy planning
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Imaging Investigations (not radiation) — Pre-hormone therapy MRI scans will be performed as an adjunct to the patients' staging MRI scan; post hormone MRI will be done wholly for research purposes.
Other: Other — Insertion of gold seeds into prostate for image registration.

SUMMARY:
To determine if functional MRI methods will aid planning of a radiation dose boost within the prostate in patients with prostate cancer potentially improving safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Hormone therapy naive patients planned to be treated by radical radiotherapy after 3-6 months of androgen suppression
* Patients with low-high risk histologically confirmed localised disease are eligible, with WHO performance status 0-1.

Exclusion Criteria:

* Patients unsuitable for functional MRI of the prostate or gold seed fiducial marker insertion (e.g. patients unable to tolerate endorectal MRI examination).
* No prior pelvic radiotherapy or radical prostatectomy, previous androgen therapy, patients unsuitable for radical radiotherapy, life expectancy <10 years, previous active malignancy within last 5 years, co-morbid conditions likely to impact on the advisability of radical radiotherapy, full anticoagulation, other exclusions to MRI (e.g. hip prosthesis or fixation, claustrophobia, ferromagnetic implants).

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of dose distributions produced by rival radiotherapy plans judged using radiobiological model predictions of Tumour Control Probability (TCP) and Normal Tissue Complication Probability (NTCP).

SECONDARY OUTCOMES:
Comparison of reproducibility of registration algorithms for mapping functional MR data acquired before hormone therapy to MR anatomical data acquired after hormone therapy and prior to radiotherapy.
Comparison of reproducibility of registration of functional and MR data with computed tomography (CT) data using gold seed registration, assessing reproducibility and positioning issues.
Comparison of image quality, registration reproducibility and gland distortion of internal and external imaging coils for MRI image acquisition and registration of the prostate.
Comparison of dose distributions produced by rival radiotherapy plans judged using three standard dose-volume constraints for targets and normal tissues and careful examination of the 3D dose distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nandita deSouza, Principal Investigator — CRUK Clinical Magnetic Resonance Research Group
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom